CLINICAL TRIAL: NCT05158101
Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Exosome Intranasal Instillations for the Treatment of Stroke
Brief Title: Safety of Cultured Allogeneic Adult Umbilical Cord Derived Mesenchymal Stem Cell Exosome Intranasal Instillations for Stroke
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Foundation for Orthopaedics and Regenerative Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ATG-2-MSC-011
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: Stroke; stem cell treatment
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (AlloEx) (Experimental): Intranasal instillations of 4 CCs of AlloEx between both nasal cavaties, which is approximately 800 billion exosomes in total. Second dose of 4 CCs to be receive the following day.
  Interventions: Biological: AlloEx

INTERVENTIONS:
Biological: AlloEx — cultured allogeneic adult umbilical cord derived mesenchymal stem cell exosomes

SUMMARY:
This trial will study the safety and efficacy of intranasal instillation of cultured allogeneic adult umbilical cord derived mesenchymal stem cell exosomes for the treatment of Stroke

DETAILED DESCRIPTION:
This patient funded trial aims to study the safety and efficacy of intranasal instillation of cultured allogeneic adult umbilical cord derived mesenchymal stem cell (UC-MSC) exosomes for the treatment of Stroke. Patients will receive intranasal instillations between both nasal cavities of UC-MSC exosomes. The total dose will be 4 CC of AlloEx, approximately 800 billion exosomes, for each day. Patients will receive instillations on back-to-back days totaling 2 doses. Patients will be evaluated within one month pre treatment and at 1, 6, 12, 24, 36, and 48 months post treatment for safety and efficacy.

For patients with more severe disease an autologous Effector cells (activated lymphocytes) treatment will be utilized created from the patient's own cells obtained by apheresis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Stroke
* Understanding and willingness to sign a written informed consent document

Exclusion Criteria:

* Active infection
* Active cancer
* Chronic multisystem organ failure
* Pregnancy
* Clinically significant Abnormalities on pre-treatment laboratory evaluation
* Medical condition that would (based on the opinion of the investigator) compromise patient's safety.
* Continued drug abuse
* Pre-menopausal women not using contraception
* Previous organ transplant
* Hypersensitivity to sulfur

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Safety (adverse events) | Four year follow-up
  Clinical monitoring of possible adverse events or complications

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Prodromos, MD, Principal Investigator — The Foundation for Orthopaedics and Regenerative Medicine
Locations (2):
- Medical Surgical Associates Center, St John's, Antigua and Barbuda
- Center for Investigation in Tissue Engineering and Cellular Therapy, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No